CLINICAL TRIAL: NCT05807217
Title: A Study to Evaluate the Pharmacokinetics of Meropenem and Piperacillin in Patients With Sepsis
Brief Title: A Pharmacokinetics Study of Meropenem and Piperacillin in Patients With Sepsis
Acronym: APSOMAPIPWS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shen Ning (Other)
Responsible Party: Sponsor-Investigator, Shen Ning, Deputy Director, Department of Respiratory and Critical Care Medicine, Peking University Third Hospital
Organization: Peking University Third Hospital (Other)
Other Study IDs: DCTC-IIR 202215
Record Dates: First submitted 2023-02-06; First posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-03

CONDITIONS: Sepsis; Acute Kidney Injury
Keywords: sepsis; organic anion transporter; acute kidney injury; quantitative pharmacology; anti-infective drug
MeSH Terms: conditions — Sepsis; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood cell
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Group A: 12 patients (receiving meropenem) without acute kidney injury
- Group B: 12 patients (receiving meropenem) without renal replacement therapy for acute kidney injury
- Group C: 12 patients (receiving meropenem) with intermittent renal replacement therapy for acute kidney injury
- Group D: 4 patients (receiving meropenem) with continuous renal replacement therapy for acute kidney injury
- Group E: 4 patients (receiving piperacillin) with intermittent renal replacement therapy for acute kidney injury

SUMMARY:
This study was a single-center, open clinical study in Chinese septic patients with or without acute kidney injury. The aims of this study were to obtain the blood concentration and pharmacokinetic parameters of meropenem and piperacillin, exosome information and endogenous biomarker, and to explore the functional changes of OATs under the condition of sepsis and acute kidney injury.

DETAILED DESCRIPTION:
The target population of this study was Chinese septic patients with or without acute kidney injury, which were divided into five groups including group A of 12 patients (receiving meropenem) without acute kidney injury, group B of 12 patients (receiving meropenem) without renal replacement therapy for acute kidney injury, group C of 12 patients (receiving meropenem) with intermittent renal replacement therapy for acute kidney injury, group D of 4 patients (receiving meropenem) with continuous renal replacement therapy for acute kidney injury and group E of 4 patients (receiving piperacillin) with intermittent renal replacement therapy for acute kidney injury. All subjects who may participate in the study must sign informed consent form (if one has no capacity for civil conduct, the guardian will sign on behalf of him), and the subjects who sign informed consent form will be screened for eligibility evaluation based on the inclusion criteria. Waste blood samples (if any) obtained from blood biochemical or routine blood tests and urine (if any) were collected in all groups and residual urine volume within 24 hours was recorded. Subjects were treated with the regimens of meropenem or piperacillin on study day (D1), which were determined and implemented by the clinician according to the treatment guidelines. Medications that may affect OAT function were not allowed during the study period (evaluated and recorded by the clinician). Venous blood was collected from all subjects at 0 h predose; at 0 h, 0.5 h, 3.5 h (Q8h) or 5.5 h (Q12h) after the end of the infusion; and within 30 min before next dose. In addition to 4 mL of venous blood taken at 0 h predose, 1 mL of venous blood should be collected at every other time point. Meanwhile, information of drug combination, complications, drug susceptibility, pathogen detection, demographic data and RRT parameters (if any) were also recorded during the period of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged above 18 years old;
2. Diagnosed with sepsis or septic shock;
3. Body mass index (BMI) between 15-32 kg/m2 (male with the weight of > 45 kg and female with the weight of > 40 kg);
4. Patients should be able to understand and sign the ICF voluntarily (if one has no capacity for civil conduct, the guardian will sign on behalf of him) and comply with the research restrictions.
5. A diagnosis of AKI by the criteria of KDIGO for Group B, C, D and E;
6. The pathogenic pathogen isolated or judged by attending physician to be susceptible to meropenem or piperacillin.
7. RRT can be performed for Group C, D and E.

Exclusion Criteria:

1. Be allergic to carbapenems and other β-lactam drugs or a history of allergy to those drugs;
2. Currently diagnosed as malignant tumor;
3. Women who are pregnant or breastfeeding;
4. Receiving ECMO during RRT;
5. Patients with severe liver insufficiency (Child-Pugh grade C);
6. Patients with eGFR of < 15 mL/min/1.73 m2 and receive regular dialysis treatment;
7. A history of alcohol or drug abuse or a behavior of alcohol or drug abuse within the past six months;
8. Patients who have taken or injected probenecid, gentamicin and streptomycin within 14 days before administration;
9. Patients who have taken or injected vitamin B6 for 14 days before administration to the trial period;
10. Poor peripheral venous access or intolerance to venous blood collection;
11. Meet one of the following conditions: human immunodeficiency virus (HIV), hepatitis B virus (HBV) surface antigen positive (except C antibody was positive), hepatitis C virus (HCV) or syphilis positive;
12. Patients who had a history of kidney transplantation or nephrectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese septic patients with or without acute kidney injury
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2022-10-26 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Plasma concentration of meropenem | Baseline and within 24 hours after administration
Dialysate concentration of meropenem | One day
Plasma concentration of piperacillin | Baseline and within 24 hours after administration
Dialysate concentration of piperacillin | One day

SECONDARY OUTCOMES:
Plasma concentration of pyridoxic acid | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ning shen, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No